CLINICAL TRIAL: NCT00530426
Title: ADHERE Core II - Acute Decompensated HEart Failure REgistry
Brief Title: Heart Failure Registry
Status: Completed | Type: Observational
Sponsor: Scios, Inc. (Industry)
Other Study IDs: CR010513
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2007-10

CONDITIONS: Heart Failure, Congestive
Keywords: Heart Failure, Congestive; Registry; Acute Decompensated Heart Failure; Dyspnea
MeSH Terms: conditions — Heart Failure; Dyspnea

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
The purpose of this registry is to compile a large clinical database on the medical management of patients hospitalized with acute heart failure, using information collected from acute care hospitals across the United States.

DETAILED DESCRIPTION:
ADHERE is a phase IV, multicenter, observational, open-label registry of the management of patients treated in the hospital for acute heart failure (HF) in the United States. The target population consists of patients admitted to an acute care hospital who are treated actively for acute heart failure, where acute HF is defined as new-onset HF with decompensation; or chronic HF with decompensation. Patient eligibility is based upon the presence of an acute HF diagnosis and is not tied to the use of any specific therapeutic agent or regimen. Collect data on the episode of hospital care beginning with the point of initial care in the hospital and/or emergency department and ending with the patient's discharge, transfer out of the hospital, or in-hospital death.

N/A

ELIGIBILITY:
Inclusion Criteria:

* Received or is eligible to receive a principal hospital discharge diagnosis of HF or decompensated HF is present as determined clinically by the patient care team

Exclusion Criteria:

* Heart Failure is present as a co-morbid condition, but is not a principal focus of diagnosis or treatment during this hospitalization episode

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150000
Dates: Start 2001-09; Study Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scios, Inc. Clinical Trial, Study Director — Scios, Inc.

REFERENCES:
- [Result] Adams KF Jr, Fonarow GC, Emerman CL, LeJemtel TH, Costanzo MR, Abraham WT, Berkowitz RL, Galvao M, Horton DP; ADHERE Scientific Advisory Committee and Investigators. Characteristics and outcomes of patients hospitalized for heart failure in the United States: rationale, design, and preliminary observations from the first 100,000 cases in the Acute Decompensated Heart Failure National Registry (ADHERE). Am Heart J. 2005 Feb;149(2):209-16. doi: 10.1016/j.ahj.2004.08.005. PMID 15846257